CLINICAL TRIAL: NCT02231645
Title: Subthalamic Deep Brain Stimulation Effects on Moral and Economics Decision-making Processing in Patients With Parkinson's Disease
Brief Title: Subthalamic Deep Brain Stimulation Effects on Decision-making Processing in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Fondazione Mondino (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DBS-Parkinson
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep brain stimulation; Subthalamic nucleus; decision-making; cognition; behavior
MeSH Terms: conditions — Parkinson Disease; Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- STN DBS group (Experimental): Experimental protocol is executed in PD patients with STN DBS implant in STN DBS ON and OFF conditions
  Interventions: Device: STN DBS
- Control group (No Intervention): Experimental protocol is executed in PD patients without STN DBS implant twice without experimental variable manipulation.

INTERVENTIONS:
Device: STN DBS — The DBS device is turned on and off by the physician.
  Arms: STN DBS group

SUMMARY:
The purpose of this study is to evaluate whether subthalamic deep brain stimulation (STN DBS) can affect moral and economic decisions in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Sample

A group of patients with idiopathic PD and with bilateral STN DBS implant (experimental group) and a control group including patients with idiopathic PD and without DBS implant who are treated with dopaminergic medications will be recruited from the IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico of Milan and from the Istituto Neurologico Nazionale IRCCS Casimiro Mondino of Pavia. Patients will be selected in order to balance groups for gender, age, disease duration, cognitive and motor functions.

Decision-making computerized tasks

Moral task. The task consisted of 38 sentences divided into 13 neutral, 10 moral conflictual and 15 moral non conflictual statements. Each statement was presented in a random order for a maximum of 10 s. During this period, participants were instructed to read each sentence and to respond if they agreed or disagreed with it by pressing the "A" (agreement) or the "L" (disagreement) keys with the left or the right finger. After the key was pressed, a black screen was displayed for 1 s before the next statement appeared on the screen (Fumagalli et al., 2011).

Economics task. Pairs of stimuli (four letters from the Latin alphabet) are presented on the screen in white on a black background. To maximize gains, subjects are asked to choose a letter by pressing one of the two keyboard keys, corresponding to the stimulus on the left or right of the screen. Each choice prompts two visual feedbacks, the first displaying the money won or lost and the second indicating the total sum of money the subject was gaining. Each stimulus pair is preceded by a black screen. Six different stimulus pairs (AB, AC, AD, BC, BD, CD) are presented. Stimulus pairs comprised stimuli with the same probability to win (conflictual trials) and different probability to win (non conflictual trials). The letters "A" and "D" led to positive feedback (+60 Euros) 80% of the times and to negative feedback (-30 Euros) 20% of the times (non risky letters). "B" and "C" letters led to high positive feedback (+100 Euros) only 20% of the times and to a high negative feedback (-70 Euros) 80% (risky letters). The task is designed to reward non risky choices, so that the larger the number of non risky choices, the higher is the amount of money earned. The task comprises 102 trials, 68 non conflictual and 34 conflictual (Rosa et al., 2013).

Experimental protocol

All patients will be tested with the moral and the economics tasks during the best ON-drug medication condition. The experimental group performed the tasks in the STN DBS ON condition and in the STN DBS OFF condition. Following the end of the STN DBS ON session, the DBS devices will be turned off by the physician 30 minutes prior to the STN DBS OFF session. The order of stimulation conditions and of the versions of the task will be randomized and counterbalanced.

The control group will similarly perform the moral and the economics tasks twice with the same time intervals, without the STN DBS manipulation.

Motor, cognitive and psychological assessment. Patients will perform a short motor, cognitive and psychological assessment using the UPDRS III, the MMSE and VASs for subjective evaluation of mood, anxiety, movement difficulty and motor fatigue. VASs will be performed twice: in STN DBS ON and OFF conditions for experimental group, and in the first and the second session for the control group. UPDRS III and MMSE will be evaluated when patients from the experimental group are in STN DBS ON condition and when control patients are in the first session.

Statistical Analysis

Normality tests will be performed on behavioural data (reaction times and responses at computerized tasks, scores obtained at MMSE, UPDRS III, VASs) with One-Sample Kolmogorov-Smirnov Test.

Behavioural data obtained by the experimental group in STN DBS ON and STN DBS OFF conditions will be compared with analysis of variance (ANOVA). Also data obtained by patients from the experimental group will be compared to data obtained by the control groups.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* For experimental group: STN DBS implant occurred no less than 6 months before and with optimal stimulation parameters

Exclusion Criteria:

* Cognitive, behavioural and psychiatric symptoms

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Reaction times and responses recorded at the moral task | For the experimental group these measures are collected in ON and OFF STN DBS (30 minutes pass between the ON and OFF condition)

SECONDARY OUTCOMES:
Reaction times and responses recorded at the economics task | For the experimental group these measures are collected in ON and OFF STN DBS (30 minutes pass between the ON and OFF condition)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Priori, MD, PhD, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico